CLINICAL TRIAL: NCT02940509
Title: The Role of Ketamine and Magnesium in Post-operative Pain Control After Laparoscopic Surgery in Patients With Chronic Pelvic Pain Treated With Opioids: A Double-Blinded Randomized Control Trial.
Brief Title: Ketamine and Magnesium in Post-operative Pain Control in Patients Treated With Opioids
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in practice of medicine. There were no longer sufficient patients to enroll in the study that met criteria.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Stacey Duryea, Physician, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00006048
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Ketamine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine plus Magnesium sulfate (Active Comparator): Ketamine 0.5mg/kg IV dose with 2g magnesium IV dose
  Interventions: Drug: Ketamine plus Magnesium sulfate
- Placebo (Placebo Comparator): Normal Saline (NaCl 0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine plus Magnesium sulfate — Patients will receive 2 IV infusions:
  1. Ketamine (0.5mg/kg)
  2. Magnesium sulfate (2g)
  Arms: Ketamine plus Magnesium sulfate
Drug: Placebo — Patients will receive 2 IV infusions, both of NaCl 0.9%, as placebos for Ketamine and magnesium sulfate
  Other Names: 2 placebo infusions
  Arms: Placebo

SUMMARY:
The goal of this research proposal is to determine if the intraoperative administrative of Ketamine and Magnesium during laparoscopic gynecologic surgery improves postoperative pain in patients on chronic opioid therapy for management of chronic pelvic pain.

DETAILED DESCRIPTION:
In this randomized control trial, patients' postoperative pain scores will be assessed as scored by the Numeric Rating Score (NRS) system. Intraoperative and postoperative narcotic usage, nausea scores and patients' perception of their quality of recovery via the QoR-40 survey will also be assessed.

The use of intraoperative Ketamine and Magnesium is predicted to decrease postoperative pain in patients on chronic opioid therapy for management of chronic pelvic pain and will overall improve patients' postoperative experience.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing elective laparoscopic gynecologic surgery
2. Patients with chronic pelvic pain defined as pain that has persisted for more than 6 months in duration which is localized to the pelvis, anterior abdominal wall, lower back or buttocks and has leads to functional disability or medical care1
3. Patients requiring opioids daily for >1 month
4. Consenting adults age 18-80
5. American Society of Anesthesiologists (ASA) Physical Status classification II to ASA III

Exclusion Criteria:

1. Patient refusal
2. Chronic Kidney disease (Creatinine>2)
3. Patients treated with methadone
4. Known allergy or adverse effect of ketamine or magnesium
5. Patient unable to give informed consent
6. Patient with limited or no English fluency
7. Uncontrolled hypertension

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Post-operative pain score using the Numeric Rating Scale (NRS) | 1st 24 hours post-op
  Patient described pain level on a scale of 0-10

SECONDARY OUTCOMES:
Post-operative opioid use | 24 hours post operative
  Dilaudid and Oxycodone in mg.
Recovery Questionnaire | 3-5 days post operative
  Patient perception of quality of recovery as measured by the QoR-40 Survey
Intraoperative fentanyl use | Intraoperative
  Amount of fentanyl used intra-operatively in mcg.
Nausea Scores using PONV Impact Scale Score | 24 hours Post operative
  Patient described nausea level using 2 questions each with 4 answers with numerical value from 0-3. To calculate the PONV Impact Scale score, the numerical responses to questions 1 and 2 are added to obtain the PONV impact scale score. A PONV Impact Scale score of ≥5 defines clinically important PONV.
Length of Hospital Stay | 24 hours Post operative
  Number of days the patient was an inpatient in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Duryea, DO, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No